CLINICAL TRIAL: NCT06953453
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Inhaled Fentanyl Aerosol (25µg/Dose) in Chinese Patients With Malignant Tumors
Brief Title: A Study of Inhaled Fentanyl Aerosol in Chinese Patients With Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZK07
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Inhaled fentanyl aerosol (Experimental): Subjects will be randomly assigned (1:1) to either drug sequence
  Interventions: Drug: Inhaled Fentanyl Aerosol
- Active Comparator:Fentanyl Citrate Injection (Active Comparator): Subjects will be randomly assigned (1:1) to either drug sequence
  Interventions: Drug: Fentanyl Citrate Injection

INTERVENTIONS:
Drug: Inhaled Fentanyl Aerosol — The subjects will be randomly assigned (1:1) to either dosing sequence: in the first cycle, receive an intravenous bolus (5 seconds) of 25μg Fentanyl injection, after at least a 2-week washout period, in the second cycle, receive a single dose of 25μg Fentanyl aerosol inhaler through the Staccato delivery system; or receive the same treatment in the reverse order.
  Arms: Experimental:Inhaled fentanyl aerosol
Drug: Fentanyl Citrate Injection — The subjects will be randomly assigned (1:1) to either dosing sequence: in the first cycle, receive an intravenous bolus (5 seconds) of 25μg fentanyl injection, after at least a 2-week washout period, in the second cycle, receive a single dose of 25μg fentanyl aerosol inhaler through the Staccato delivery system; or receive the same treatment in the reverse order.
  Arms: Active Comparator:Fentanyl Citrate Injection

SUMMARY:
This study is a single-dose, open-label, 2-cycle crossover design, comparing the pharmacokinetic parameters and safety of Inhaled Fentanyl Aerosol and intravenous fentanyl injection.

DETAILED DESCRIPTION:
Consenting patients who met inclusion and exclusion criteria were allowed to enter the study. The subjects will be randomly assigned (1:1) to receive an intravenous bolus (5 seconds) of 25μg fentanyl injection in the first cycle, and after a 2-week washout period, to receive a single dose of 25μg inhaled fentanyl aerosol through the Staccato delivery system in the second cycle; or to receive the same treatment in the opposite order.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate, understand and sign the informed consent form before conducting the evaluation project;
2. Male or female subjects, aged between 18 and 55, including 18 and 55 years old;
3. Patients with malignant tumors diagnosed by histology or cytology;
4. Body Mass Index (BMI) is >21 kg/m2, but <30 kg/m2;
5. Have sufficient hematopoietic function and organ function within the last 14 days at random.

   1. The absolute neutrophil count is ≥1.5×109/L (has not received colony stimulating factor treatment within 14 days before the examination);
   2. Platelet count ≥80×109/L (without transfusion of platelets or other platelet-increasing drugs within 14 days before the examination);
   3. Hemoglobin ≥90g/L (without transfusion or treatment with other hemoglobin-increasing drugs within 7 days before the examination);
   4. Creatinine clearance rate (Ccr)≥30 ml/min, Cr≤2 times the upper limit of normal value;
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) should be ≤2.5×ULN, and for subjects with liver metastasis, it should be ≤5×ULN; total bilirubin should be ≤2 times the upper limit of normal value;
   6. Coagulation function INR≤1.5 ULN;
   7. In a non-oxygen-absorbing state, the oxygen saturation (from a pulse oximeter) is SaO2>95%; pulmonary function shows FEV1/FVC>70% and FEV1 as a percentage of the predicted value is>80%;
6. All patients must agree to take effective contraceptive measures during the study and within one month after stopping treatment. Female patients of childbearing age must have a negative blood pregnancy test before administration;
7. The ECOG performance status score is 0~1 points;

Exclusion Criteria:

1. known or suspected allergy to opioids;
2. used opioids within 14 days before the first administration, including but not limited to: codeine, dihydrocodeine, hydromorphone, oxycodone, methadone, morphine, fentanyl and pethidine (pethidine);
3. plan to receive radiotherapy and / or systemic chemotherapy within 14 days before the first administration or during the study period (except for patients who receive immune checkpoint inhibitors or targeted drug maintenance therapy that is not a CYP3A4 inhibitor / inducer and whose condition is stable);
4. within 14 days before the first administration, the patient had received any monoamine oxidase (MAO) inhibitors (such as phenelzine, isocarbazine, chlorogiline, toloxadone, moclobemide, selegiline, rasagiline, etc.); Or have used CYP3A4 inhibitors (such as indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, nefazodone, ketoconazole, telithromycin, arepitan, erythromycin, fluconazole, grapefruit, verapamil, diltiazem, cimetidine, etc.) or CYP3A4 inducers (such as phenobarbital, carbamazepine, efavirenz, glucocorticoids, modafinil, nevirapine, oxcarbazepine, phenytoin, pioglitazone, rifabutin, rifampicin);
5. have participated in other clinical studies or received surgical treatment within 30 days before the screening period, or have surgery plans during the study period;
6. subjects who smoked more than 10 cigarettes / day within 3 months before the screening period;
7. subjects with a history of drug or alcohol dependence or abuse within 2 years before the screening period;
8. subjects often eat food rich in xanthine (such as drinking more than 5 cups of coffee or food containing the same amount of xanthine every day);
9. subjects with hypotension (systolic blood pressure <90 mmHg, or diastolic blood pressure <60 mmHg) or uncontrollable hypertension (refers to systolic blood pressure ≥ 160 mmHg, and / or diastolic blood pressure ≥ 100 mmHg after standard treatment);
10. After antiviral treatment, HBV DNA>500 IU/mL or>2500 copies/mL; HCV-RNA positive; Positive for human immunodeficiency virus antibodies; Or positive for syphilis antibodies;
11. subjects with positive alcohol test or urine test at any visit of the study;
12. subjects with an expected survival time of <1 year;
13. subjects with clinically significant ECG abnormalities during screening;
14. subjects with a history of lung diseases (asthma, bronchitis, bronchospasm, emphysema, interstitial lung disease, pulmonary fibrosis, etc., excluding lung malignancies);
15. subjects with history of unstable angina pectoris, syncope, coronary artery disease, myocardial infarction, congestive heart failure (CHF), stroke, transient ischemic attack (TIA) or major neurological diseases;
16. presence of meningeal metastasis or CNS metastasis requiring clinical intervention or malignancy related epilepsy;
17. women of childbearing age or lactating women with positive blood and urine pregnancy tests;
18. the investigator believes that any other situation that may affect the subject's provision of informed consent or compliance with the trial protocol, or the subject's participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Cmax | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Peak Concentration
Tmax | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Time to Maximum Concentration
Ke | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Terminal Elimination Rate
T1/2 | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Terminal elimination half-life
CL/F | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Apparent Clearance (CL/F)
AUC_last | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Area Under the Concentration-Time Curve from Time Zero to the Last Quantifiable Concentration
AUC_inf | Before administration (within 30 minutes), 15 seconds , 30 seconds, 45 seconds, 90 seconds, 3 minutes, 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 18 hours after administration
  Area Under the Concentration-Time Curve from Time Zero to Infinity

SECONDARY OUTCOMES:
Pupil diameter | Pupil measurements were taken before administration, and at 1, 2, 3, 5 , 10 , 30minutes , and 1, 2, 4, 8, 12 and 18hours after drug administration.
  Measure the pupil diameter using a pupillometer.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Hu, doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (2):
- China (2):
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No